CLINICAL TRIAL: NCT04115267
Title: Attribution of Toxicities Due to Radiotherapy and Immuno-Biological Therapies - Registry
Brief Title: Attribution of Toxicities Due to Radiotherapy and Immuno-Biological Therapies
Acronym: AtTRIBut
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 19.065
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Cancer; Radiotherapy Side Effect
Keywords: Combined effect; Registry; Side effects; Patient reported outcome; Cancer
MeSH Terms: conditions — Neoplasms; Radiation Injuries | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Combined modality: Patients receiving radiotherapy and a molecular agent for the treatment of cancer
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Combined modality
  Other Names: Anti-neoplastic Molecular Agent

SUMMARY:
Every year, new molecular agents enter the market with more and more patients receiving these treatments, especially in the metastatic setting. These molecular agents could correspond to immunotherapy and modulators of signaling pathways. More than 50% of cancer patients will receive radiation therapy during the course of their illness, including radiotherapy aimed a palliating symptoms secondary to metastatic diseases. Therefore, there will be an increasing number of patients who will be receiving radiotherapy while they are still receiving molecular agents. A better understanding of the interaction of these two treatment modalities is needed.

DETAILED DESCRIPTION:
Every year, new molecular agents enter the market with more and more patients receiving these treatments, especially in the metastatic setting. These molecular agents could correspond to immunotherapy and modulators of signaling pathways. More than 50% of cancer patients will receive radiation therapy during the course of their illness, including radiotherapy aimed a palliating symptoms secondary to metastatic diseases. Therefore, there will be an increasing number of patients who will be receiving radiotherapy while they are still receiving molecular agents. A better understanding of the interaction of these two treatment modalities is needed.

It is within this context that this registry was set up to gather information from physicians and patients treated with molecular agents and radiation therapy. The information being collected include diagnosis, doses received, type of targeted therapy, side effects, etc. Through this registry, we wish to determine whether there are more Grade 3 or above side effects than what is reported in the literature for these treatment modalities, when given alone or in combination. Participating patients will also describe their perceived side effects and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Consent to be part of the AtTRIBut registry
* Prior histological diagnosis of primary cancer.
* If the patient has metastatic disease, there must be radiological or pathological evidence of metastasis
* Age> 18 years
* Receiving a molecular therapy
* Indicated to receive radiotherapy
* Radiation therapy can be administered using 3D conventional, IMRT or SBRT techniques.

Exclusion Criteria:

• Refusal or inability to receive radiotherapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients planned to be treated with radiotherapy and who are receiving a targeted therapy, including immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2019-09-13 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with severe side effects | 1 year
  CTCAE V5 Grade 3-5 toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Philip Wong, MD, Principal Investigator — CHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No